CLINICAL TRIAL: NCT02112409
Title: Autologous Blood Transfusion Technique in Idiopathic Scoliosis Surgery - a Comparison Between Intraoperative Cell Salvage With Hemodilution Techniques Versus Cell Salvage Technique Alone
Brief Title: Intraoperative Cell Salvage and Hemodilution Technique in Scoliosis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 201312-0621
Record Dates: First submitted 2014-04-05; First posted 2014-04-14 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adolescent idiopathic scoliosis; scoliosis corrective surgery; autologous blood transfusion; cell salvage; acute normovolemic hemodilution; hemoglobin level

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cell salvage and hemodilution technique (Experimental): cell salvage technique throughout scoliosis corrective surgery; Acute normovolemic hemodilution technique commenced after induction of anaesthesia and prior the starting of surgery.
  Interventions: Procedure: cell salvage technique; Procedure: acute normovolemic hemodilution
- cell salvage (Active Comparator): cell salvage technique throughout scoliosis corrective surgery
  Interventions: Procedure: cell salvage technique

INTERVENTIONS:
Procedure: cell salvage technique — blood from the surgical field is collected, anti-coagulated, filtered, centrifuged, washed and re-suspended in saline to produce autologous blood with a resultant haematocrit of 50-80% for transfusion back to the patient using specific cell saver device
  Other Names: intraoperative blood salvage using cell saver
Procedure: acute normovolemic hemodilution — Removal of 500ml whole blood from the patient after induction of anesthesia, with restoration of blood volume with acellular fluid using equivolume of 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride (voluven) to maintain isovolemia
  Other Names: intraoperative hemodilution technique
  Arms: cell salvage and hemodilution technique

SUMMARY:
Surgical correction of scoliosis with instrumentation carries significant blood loss and needs for blood transfusion with its inherent risk and cost. In recent years, there is an increased interest in utilizing autologous blood as part of perioperative blood conservation strategy.

The foremost mechanical methods of perioperative conservation of red blood cells including intraoperative cell salvage (ICS) and acute normovolemic hemodilution (ANH). They should be considered in all cases where significant blood loss (>1000 ml) or >20% estimated blood volume is expected, in patients with multiple antibodies or rare blood types and those who refuse allogenic blood products.

Literature search has revealed that both cell salvage method and ANH utilized in elective surgeries are capable of minimizing allogenic blood transfusion respectively. Surgeries which are of significant relevance are aortic surgery, cardiac surgery and arthroplasty orthopaedic surgery. Combining the above two techniques such as in ATIS trial 2002 also shows that it is safe and significantly reduced allogenic blood requirements in aortic surgery. However till date, there is still lack of strong evidence that autologous blood transfusion technique is beneficial for scoliosis surgery in reducing allogenic blood transfusion.

Hypothesis:

The investigators hypothesize that the addition of ANH to ICS would confer additional benefit than using cell saver alone. By combining cell saver with hemodilution technique, the difference between pre-operative and post-operative Hemoglobin level will be smaller than using cell saver technique alone, hence minimizing the variation in perioperative Hemoglobin level - a predictor of allogenic blood transfusion.

DETAILED DESCRIPTION:
Patients who meet the inclusion criteria are enrolled in the study. They are assigned to 2 arms of study group using concealed allocation method. A computerized random-number generator will be used to formulate an allocation schedule. Group A will receive cell salvage and acute normovolemic hemodilution during operation; Group B will only receive cell salvage as sole autologous transfusion strategy.

Members of the research team should attend all operations and record all data. Anaesthetic technique including drugs usage, equipments and monitoring devices are standardized as per protocol. Intraoperative fluid management is recorded in details.

All patients enrolled in the study (group A and B) underwent cell saver technique during surgery using Cell Saver® 5+ autologous blood recovery system-Haemonetics devices. All patients allocated in group A also received additional acute normovolemic hemodilution (ANH) after induction of anaesthesia. As a standardization measure, before starting skin incision, 500ml blood will be collected from the radial artery to a standard blood collection bag and stored as CPD blood at ambient temperature. Simultaneously, 500ml Voluven® (6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride) will be infused through a peripheral vein.

All autologous blood will be re-infused back to patient at surgery completion or within 6 hours of withdrawal. Autologous blood will be given to patient during surgery at any point if there are 30% or more body blood volume loss.

Allogenic blood will be administered when the intraoperative hemoglobin concentration fell below 8g/dl despite completion of autologous blood transfusion or when autologous blood not available; adequate volume correction by mean of collected autologous blood and crystalloid fluid administration, or when presence of ischemic electrocardiogram changes (2mV ST segment elevation or depression on 3 leads monitoring); persistent hypotension or tachycardia >20% from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Elective single stage posterior spinal fusion for scoliosis corrective surgery
* Diagnosis of idiopathic scoliosis
* Age >10 and <25
* ASA I or II
* Preoperative Hemoglobin > 10 g/dL
* Preoperative Platelet > 150,000/L
* Clinically fit for surgery
* Written informed consent

Exclusion Criteria:

* Patient's refusal of homologous blood
* Hematological disorder rendering either transfusion technique inappropriate
* Patients who received anticoagulants and antiplatelets perioperatively
* Severe cardiac disease (Aortic stenosis or cardiac ejection fraction <40%; Myocardial infarction in the previous 6 Months; Myocardial ischaemia on resting Electrocardiogram)
* Severe pulmonary disease (FEV1 50% predicted, PaO2 9 kpa on air)
* Preoperative creatinine >200 mmol/L
* AST >100 IU/L

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difference in pre-operative and post-operative hemoglobin level | at 0 hour and 24 hour post-operation
  Laboratory testing for hemoglobin level will be carry out at 0 hour and 24 hour post-operation.

SECONDARY OUTCOMES:
Perioperative requirement of allogenic blood transfusion | one week post-operation
  participants (patients) will be followed for the duration of hospital stay, an expected average of one week.

CONTACTS AND LOCATIONS:
Overall Officials: M Shahnaz Hasan, MBBS, MAnaes, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia